CLINICAL TRIAL: NCT06672510
Title: Safety and Effectiveness of the Akura Thrombectomy System for Use in the Removal of Emboli From the Pulmonary Arteries in Treating Acute Pulmonary Embolism (PE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akura Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-60006
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Patients with Acute Pulmonary Embolism (Experimental): Patients undergoing mechanical thrombectomy for acute pulmonary embolism.
  Interventions: Device: ATC

INTERVENTIONS:
Device: ATC — The ATC System is designed to mechanically remove emboli and restore blood flow through the pulmonary arteries in patients experiencing acute P

SUMMARY:
This study is a prospective, single-arm, interventional, multicenter study to evaluate the safety and effectiveness of percutaneous mechanical thrombectomy using the Akura Thrombectomy System in subjects with acute pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years of age or older and deemed medically eligible for interventional procedure, per institutional guidelines and clinical judgement
* Clinical signs, symptoms and presentation consistent with acute PE
* PE symptom duration ≤ 14 days
* CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery)
* CTA evidence of RV/LV ratio of ≥ 0.9 (NOTE: Enrollment qualification assessment is based on the Investigator's interpretation of RV/LV ratio at baseline)
* Systolic BP ≥ 90 mmHg (initial SBP may be < 90 mmHg but ≥ 80 mmHg if the pressure recovers with volume resuscitation)
* Stable HR < 130 BPM prior to the procedure

Exclusion Criteria:

* Prior PE <180 days from index procedure
* Thrombolytic use within 30 days prior to baseline CTA
* Pulmonary hypertension with peak pulmonary arterial pressure (PAP) > 70 mmHg by right heart catheterization
* Vasopressor requirement after fluids to keep pressure at ≥ 90 mmHg
* FiO2 requirement > 40% or > 6 LPM (to keep oxygen saturation > 90%)
* Hematocrit < 28% (Note: hematocrit required within 6 hrs. of index procedure)
* Platelets < 100,000/μL
* eGFR <30 ml/min per 1.73 m2
* International normalized ratio (INR) > 3
* Major trauma injury severity score (ISS) > 15
* Presence of intracardiac lead in right ventricle or atrium placed ≤ 6 months of enrollment
* Cardiovascular or pulmonary surgery within the last 7 days
* Actively progressing cancer treated by chemotherapeutics
* Known bleeding diathesis or coagulation disorder
* Left bundle branch block
* History of severe or chronic pulmonary arterial hypertension
* History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
* History of uncompensated heart failure.
* History of underlying lung disease that is oxygen dependent
* History of chest irradiation
* History of heparin-induced thrombocytopenia (HIT)
* Contraindication to systemic or therapeutic doses of anticoagulants
* Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
* Known residual iliac deep vein thrombosis (DVT), inferior vena cava (IVC) clot or clot in transit (right atrium and/or right ventricle)
* CTA imaging or other evidence that suggest, in the opinion of the investigator, the Subject is not appropriate for mechanical thrombectomy intervention (e.g. inability to navigate to target location, predominantly chronic clot or non-clot embolus)
* Life expectancy < 90 days, as determined by investigator (e.g., stage 4 cancer, frailty or severe COVID infections)
* Female who is pregnant or nursing
* Current participation in another investigational drug or device treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 48 hours
  Change in RV/LV ratio from baseline
Safety: Composite of Major Adverse Device-Related Events | 48 hours post index procedure
  Device-related major bleeding at access, device-related death, clinical deterioration, pulmonary vascular injury or cardiac injury

SECONDARY OUTCOMES:
Safety: Composite of Major Adverse Events | 30 days post index procedure
  Assessment of major adverse events through 30 day follow-up

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Advanced Heart & Vein (ClinRe-001-001), Thornton, Colorado
  - Hartford Healthcare, Hartford, Connecticut
  - Manatee Hospital / Nova Clinical Research Center, Bradenton, Florida
  - Jacksonville Memorial (HCA), Jacksonville, Florida
  - Tallahasse Memorial Hospital, Tallahassee, Florida
  - Centracare Heart & Vascular Center, Saint Cloud, Minnesota
  - Columbia University Medical Center, New York, New York
  - Cumc/Nyph, New York, New York
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - Methodist San Antonio (HCA), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No